CLINICAL TRIAL: NCT07375693
Title: Effect of Melatonin on Oxidative Stress Parameters in Levodopa-Treated Parkinson's Disease Patients: A Randomized, Double-Blind, Placebo-Controlled Trial.
Brief Title: Effect of Melatonin on Oxidative Stress Parameters in Levodopa-Treated Parkinson's Disease Patients
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Bangladesh Medical University (Other)
Responsible Party: Principal Investigator, Dr. Farzana Akter, principal investigator, Bangladesh Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: BSMMU/2025/4251
Record Dates: First submitted 2025-12-10; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-05

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): participants received Melatonin 10 mg orally 1 tab daily 30 min before bedtime for 12 weeks
  Interventions: Drug: MELATONIN (MELATL07959)
- placebo group (Placebo Comparator): participants received placebo for 12 weeks
  Interventions: Drug: MELATONIN (MELATL07959)

INTERVENTIONS:
Drug: MELATONIN (MELATL07959) — melatonin 10 mg orally 1 tab daily 30 min before bedtime for 12 weeks
  Other Names: Tab. melatonin 10 mg

SUMMARY:
In Bangladesh Melatonin is currently used for insomnia. Its potential therapeutic benefits beyond sleep regulation. This study aimss to evaluate the effects of melatonin supplementation on oxidative stress markers, neuroinflammation and clinical outcomes in patients with Parkinson's disease. The main question it aims to answer:

In patients with Parkinson's disease receiving levodopa, does melatonin supplementation, compared to levodopa treatment alone, improve the symptoms of PD over a 12 week of period.

Participants will:

Take Melatonin 10mg or placebo everyday for 3 months at night 30minutes before bedtime. Visit the clinic once every 6 weeks for checkups and tests keep a diary of their symptoms,UPDRS score. At the end of 12 weeks will reaper hs-CRP, MDA and GSH.

DETAILED DESCRIPTION:
This research will be conducted in the Department of Pharmacology in collaboration with the Department of Neurology, at Bangabandhu Sheikh Mujib Medical University.

Patients will be recruited from the PD clinic, OPD at Department of Neurology.

Study procedure:

Mild to moderate Parkinson's disease patients receiving levodopa according to Hoehn and Yahr staging, stage -I, II, Ill will be selected from the outpatient department of the Neurology, BSMMU. The objective, nature, purpose and potential risk of all the procedures used for the study will be explained in detail to each subject, with a cordial attitude emphasizing the benefits he/she might obtain from this study.

Total of 70 patients will be assessed. Informed written consent from each patient will be taken in a prescribed form. Then demographic Information, address, mobile number, and medical history will be recorded in a preformed data schedule. For giving intervention, patients will be divided into two groups group A and group B by randomization. A total of 70 patients will be randomized, for (group A n=35) and Group B (n=35). At baseline, the MDS-UPDRS score will be evaluated by the present researcher and 6 ml blood will be collected for the baseline measurement of MDA, GSH, and hs-CRP levels. Then patients will be assigned to the respective groups. Tab. Melatonin 10mg/day (1 tablet 1 hour before bedtime) will be given to the patient of group A for 12 weeks and Tab. Placebo will be given to the patient of group B for 12 weeks. Regular medicine intake will be confirmed by talking to the patients or the care giver over the telephone and from the compliance sheet of the patients. The disease severity will be assessed by MDS-UPDRS(Part-II) score at the end of the12 weeks treatment. 6 ml blood will be collected to measure MDA, GSH and hs-CRP levels at the end of the 12 weeks of treatment. Patients will be asked to report any unwanted effects of the medicine like excessive fatigue, depression and weight loss given during the study.

First, the suspected PD patients will be evaluated by a neurologist in the neurology department. The proposed study will be conducted among outdoor patients with Parkinson's disease in the PD clinic, will be made clinically using to scale by an expert neurologist following inclusion and exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* diagnosesd Parkinson's disease patients taking levodopa
* mild to moderate PD pt according to Hohen and Yahr staging, stage-I,II,III
* age:>45 years
* both male and female

Exclusion Criteria:

* secondary causes of PD
* Prior stereotactic surgery for PD
* suffering from active malignancy
* known hypersensitivity to melatonin
* Patients taking anticonvulsants, OCP, DMARD
* pt with autoimmune disease
* pregnancy or lactating mother
* has any clinically significant medical condition that could interfere with the subject's ability to safely participate in the study or to be followed

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-02-17 (Estimated); Primary Completion 2026-08-23 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
effect of melatonin 2) Antioxidant marker erythrocyte glutathione (GSH) This study involves a comparison of MDA and GSH levels between the control and intervention groups at baseline and after 12 weeks. | 0 week and 12 weeks
  To evaluate the effect of melatonin on oxidative stress, neuroinflammation, and the improvement of symptoms in levodopa-treated PD patients.

SECONDARY OUTCOMES:
the level of oxidative stress markers | 0 week and 12 weeks
  To compare the level of oxidative stress markers including MDA and GSH in levodopa-treated PD patients
the serum hs-CRP level | 0 weeks and12 weeks
  To estimate and compare the serum hs-CRP level in levodopa-treated PD patients
using the MDS-UPDRS (Part-II) | 0 week and 12 weeks
  To assess and compare the severity score of motor activity in Levodopa treated PD patients

CONTACTS AND LOCATIONS:
Overall Officials: Farzana Akter, MBBS, Principal Investigator — Bangladesh Medical University
Locations (1):
- Bangladesh medical university, Dhaka, Dhaka Division, Bangladesh

IPD SHARING:
Plan to Share IPD: No